CLINICAL TRIAL: NCT04025086
Title: Perioperative Goal Directed Therapy (PGDT) in Spinal Surgery in the Prone Position: Optimization of Fluid Therapy, Haemodynamic Impact and on Post-operative Complications
Brief Title: Perioperative Goal Directed Therapy (PGDT) in Spinal Surgery in the Prone Position
Acronym: PGDT
Status: Completed | Type: Observational
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Marinella Astuto, Full Professor, University of Catania
Other Study IDs: 52/2018/PO
Record Dates: First submitted 2019-07-15; First posted 2019-07-18 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Intraoperative Hypotension; Pulmonary Complication; Cardiovascular Complication
Keywords: Spinal Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: 44 patient undergoing spinal surgery in prone position at "Gaspare Rodolico Presidium", in which the new "Perioperative Goal Directed Therapy" protocol has been used
- Control group: 44 patients who underwent spinal surgery in the period January 2016 - December 2017, in which was not used a Perioperative Goal Directed Therapy approach but a classical hemodynamic monitoring, according to the recommendations of good clinical practice and the international guidelines.

SUMMARY:
This study aims at evaluating if a specific protocol, that can be framed in the innovative concept of Perioperative Goal Directed Therapy (PGDT), based on the evaluation of the Stroke Volume Variation (SVV) - a parameter deriving from the adoption of a minimally invasive advanced hemodynamic monitoring technology with a special sensor called FloTrac® (Edwards) or of a non-invasive monitoring system with the Clearsight® sensor (Edwards) - is able to guarantee a greater precision in the intraoperative management of patients undergoing spinal surgery in prone position.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-80 years
* American Society of Anesthesiologists(ASA) Classification I-II-III
* Minor and major spinal surgery
* Prone position
* Sinus rhythm
* Absence of atrial fibrillation. or severe arrhythmia
* Informed consent

Exclusion Criteria:

* Absence of informed consent
* Age less than 18 or older than 80 years
* Cardiac rhythm abnormalities: atrial fibrillation and / or severe arrhythmia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 44 Patients undergoing spinal surgery in prone position at "Gaspare Rodolico Presidium" of Policlinico-Vittorio Emanuele University Hospital of Catania, in which a specific protocol, that can be framed in the innovative concept of Perioperative Goal Directed Therapy (PGDT), based on the evaluation of the Stroke Volume Variation (SVV) by using a minimally invasive advanced hemodynamic monitoring technology with a special sensor called FloTrac® (Edwards) o a non-invasive monitoring system with Clearsight® sensor (Edwards), is used.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Frequency rate of early post-operative complications | 7 days

SECONDARY OUTCOMES:
Comparison between the two commonly adopted anesthetic techniques (totally intravenous anesthesia (TIVA / TCI) or balanced anesthesia) in terms of intraoperative management of the patient and post-operative complication | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Gaspare Rodolico Presidium - University Hospital Policlinico-Vittorio Emanuele, Catania, Sicily, Italy